CLINICAL TRIAL: NCT03811002
Title: Limited Stage Small Cell Lung Cancer (LS-SCLC): A Phase III Randomized Study of Chemoradiation Versus Chemoradiation Plus Atezolizumab
Brief Title: Testing the Addition of a New Immunotherapy Drug, Atezolizumab (MPDL3280A), to the Usual Chemoradiation (CRT) Therapy Treatment for Limited Stage Small Cell Lung Cancer (LS-SCLC)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-00178; NCI-2019-00178 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-LU005 (Other: NRG Oncology); NRG-LU005 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2019-01-18; First posted 2019-01-22 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-08

CONDITIONS: Limited Stage Lung Small Cell Carcinoma; Stage I Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiotherapy, Conformal; atezolizumab; Specimen Handling; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Etoposide; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (chemotherapy, radiation therapy) (Active Comparator): Patients receive etoposide IV on days 1-3 and cisplatin IV or carboplatin IV on day 1. Cycles repeat every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo 3D-CRT or IMRT BID for approximately 3 weeks or QD for approximately 6-7 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo blood specimen collection throughout the trial.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide; Radiation: Intensity-Modulated Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (chemotherapy, radiation therapy, atezolizumab) (Experimental): Patients receive treatment as in Arm I. Patients also receive atezolizumab IV over 30-60 minutes on day 1 or 2 of each chemotherapy cycle. Cycles repeat every 3 weeks for 17 cycles (1 year) in the absence of disease progression or unacceptable toxicity. Patients undergo blood specimen collection throughout the trial.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Atezolizumab; Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide; Radiation: Intensity-Modulated Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3D-CRT
  Other Names: 3-dimensional radiation therapy; 3D Conformal; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D radiotherapy; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation, 3D Conformal; Three dimensional external beam radiation therapy (procedure)
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
  Arms: Arm II (chemotherapy, radiation therapy, atezolizumab)
Procedure: Biospecimen Collection — Correlative studies
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial studies how well chemotherapy and radiation therapy (chemoradiation) with or without atezolizumab works in treating patients with limited stage small cell lung cancer. Drugs used in chemotherapy, such as etoposide, cisplatin, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving chemoradiation with or without atezolizumab may work better in treating patients with limited stage small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare overall survival (OS) for patients with LS-SCLC treated with chemoradiation +/- atezolizumab.

SECONDARY OBJECTIVES:

I. To compare progression free survival (PFS) for patients with limited stage small cell lung cancer (LS-SCLC) treated with chemoradiation +/- atezolizumab.

II. To determine overall response rate (ORR), rates of local control, and distant metastases free survival with chemoradiation +/- atezolizumab.

III. To characterize immune mediated and non-immune mediated toxicity from chemoradiotherapy plus atezolizumab.

IV. To compare quality of life, as measured by the Functional Assessment of Cancer Therapy-Trial Outcome Index (FACT-TOI), for patients undergoing chemoradiation +/- atezolizumab.

V. To evaluate the quality-adjusted survival, using scores from the 5-level EuroQol 5-dimensional questionnaire (EQ-5D-5L), of chemoradiation +/- atezolizumab for patients with LS-SCLC.

VI. To characterize fatigue, as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS), following chemoradiation +/- atezolizumab.

VII. To determine the association of small cell lung cancer (SCLC) molecular subtypes with clinical outcomes.

EXPLORATORY OBJECTIVES:

I. To collect biospecimens at baseline, day 1 and 3 months after the end of chemoradiotherapy, to allow for future analyses.

II. To characterize patient-reported symptomatic toxicities measured by the Patient-Reported Outcomes - Common Terminology Criteria for Adverse Events (PRO-CTCAE).

III. To characterize the concordance between tumor and circulating cell-free deoxyribonucleic acid (cfDNA)-determined molecular subtypes.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive etoposide intravenously (IV) on days 1-3 and cisplatin IV or carboplatin IV on day 1. Cycles repeat every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo three-dimensional conformal radiation therapy (3D-CRT) or intensity-modulated radiation therapy (IMRT) twice daily (BID) for approximately 3 weeks or once daily (QD) for approximately 6-7 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo blood specimen collection throughout the trial.

ARM II: Patients receive treatment as in Arm I. Patients also receive atezolizumab IV over 30-60 minutes on day 1 or 2 of each chemotherapy cycle. Cycles repeat every 3 weeks for 17 cycles (1 year) in the absence of disease progression or unacceptable toxicity. Patients undergo blood specimen collection throughout the trial.

After completion of study treatment, patients are followed up every 3 months for 2 years, then every 6 months for 3 years, then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of limited stage small cell lung cancer (Stage Tx, T1-T4, N0-3, M0, American Joint Committee on Cancer [AJCC] staging, 8th edition [Ed.]), within 60 days prior to registration
* Patients must have received one cycle of platinum/etoposide chemotherapy pre-registration (prior to study entry). Study registration must be within 21 days from day 1 of the pre-registration cycle of chemotherapy.
* Patients must have had measurable disease (per Response Evaluation Criteria in Solid Tumors [RECIST], version 1.1) prior to the required pre-registration cycle of platinum/etoposide chemotherapy
* Minimal staging requirements include:

  * History/physical examination within 30 days prior to registration
  * Positron emission tomography (PET)/computed tomography (CT) scan for staging within 60 days prior to registration
  * CT chest and CT abdomen with IV contrast (unless contraindicated based on kidney function) within 60 days prior to registration; magnetic resonance imaging (MRI) abdomen with IV contrast allowed in place of CT abdomen

    * Note: If contrast allergy exists, premedication per institutional guidelines should be performed prior to obtaining CT with contrast. The only exception to this is a documented life-threatening allergy
  * MRI scan of the brain with contrast (preferred) or CT scan of the brain with contrast (allowable if there is a contraindication with MRI with contrast) within 30 days prior to registration
* Age >= 18
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 within 30 days prior to registration
* Absolute neutrophil count (ANC) >= 1,500/cells/mm^3 (prior to pre-registration cycle)
* Platelet count >= 100,000 cells/mm^3 (prior to pre-registration cycle)
* Hemoglobin >= 9 g/dL (prior to pre-registration cycle)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (prior to pre-registration cycle)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.0 x ULN (prior to pre-registration cycle)
* Adequate renal function within 30 days prior to registration defined as follows: Creatinine clearance >= 30 mL/min by the Cockcroft-Gault (C-G) equation
* Patients presenting with a pleural effusion will be eligible if thoracentesis is cytologically negative and non-bloody or if pleural fluid is too small a volume to effectively sample by thoracentesis and does not show increased metabolic activity on CT/PET imaging
* Negative serum pregnancy test within 14 days of registration for pre-menopausal women of childbearing potential
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry
* Hepatitis B/C testing prior to enrollment for patients that have not been tested before. Note: This is required even if the patient has never shown or had symptoms of hepatitis
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial

Exclusion Criteria:

* Definitive clinical or radiologic evidence of metastatic disease
* Definitive surgical resection of small cell lung cancer
* Prior invasive malignancy (except non-melanomatous skin cancer, localized prostate cancer, or any early stage cancer treated with curative intent resection) unless disease free for a minimum of 2 years (carcinoma in situ of the breast, oral cavity, or cervix are all permissible)
* More than 1 cycle of prior platinum-based chemotherapy for SCLC prior to enrollment; note that prior chemotherapy for a different cancer is allowable
* Any prior atezolizumab or other immunotherapy agent
* Prior radiotherapy to the lungs or mediastinum that would result in clinically significant overlap of radiation therapy fields; prior tangent fields for breast cancer with minimal overlap with target volumes are allowed per approval of study principal investigators (PIs)
* Patients with cytologically positive pleural or pericardial fluid are not eligible
* An active, known or suspected autoimmune disease. Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* History of allogeneic organ transplant
* History of primary immunodeficiency
* Severe, active co-morbidity defined as follows:

  * Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, cirrhosis, fatty liver, and inherited liver disease
  * Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
  * Active tuberculosis
  * Active hepatitis B (chronic or acute) or hepatitis C infection. Note that if hepatitis status is unknown, hepatitis B/C testing is required

    * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg]) test, a positive anti-HBc (antibody to hepatitis B core antigen), and a negative viral deoxyribonucleic acid (DNA) test (only obtained if HBsAg is found positive) are eligible
    * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA). (The HCV RNA test must be performed for patients who have a positive HCV antibody test.)
  * Known immunosuppressive disease, for example history of bone marrow transplant or chronic lymphocytic leukemia (CLL)
  * Chronic obstructive pulmonary disease (COPD) requiring chronic oral steroid therapy of > 10 mg prednisone daily or equivalent at the time of registration. Inhaled corticosteroids are not exclusionary
  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 3 months
  * Transmural myocardial infarction within the last 3 months
  * Clinically significant interstitial lung disease
* A condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception for the duration of study treatment and for 150 days after the last dose of study drug (Arm 2); this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2024-04-21 (Actual); Study Completion 2029-02-21 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin A Higgins, Principal Investigator — NRG Oncology
Locations (543):
- United States (533):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sutter Auburn Faith Hospital, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - GenesisCare USA - Aventura FP, Aventura, Florida
  - GenesisCare USA - Aventura, Aventura, Florida
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Regional Cancer Center-Lee Memorial Health System, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - The Watson Clinic, Lakeland, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Piedmont Newnan Hospital, Newnan, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Alton Memorial Hospital, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Community Cancer Center East, Indianapolis, Indiana
  - Community Cancer Center South, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Baptist Health Floyd, New Albany, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Saint Elizabeth Healthcare Edgewood, Edgewood, Kentucky
  - Baptist Health Hardin, Elizabethtown, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Norton Audubon Hospital and Medical Campus, Louisville, Kentucky
  - Norton Brownsboro Hospital and Medical Campus, Louisville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Covington, Covington, Louisiana
  - Mary Bird Perkins Cancer Center - Houma, Houma, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - MaineHealth Coastal Cancer Treatment Center, Bath, Maine
  - MaineHealth Waldo Hospital, Belfast, Maine
  - MaineHealth Maine Medical Center - Biddeford, Biddeford, Maine
  - MaineHealth Stephens Hospital, Norway, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth Cancer Care and IV Therapy - Sanford, Sanford, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute at Boston Medical Center - Brighton, Brighton, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Michigan Healthcare Professionals Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan Healthcare Professionals Farmington, Farmington Hills, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - Mid-Michigan Physicians-Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Michigan Healthcare Professionals Macomb, Macomb, Michigan
  - Michigan Healthcare Professionals Madison Heights, Madison Heights, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Michigan Healthcare Professionals Troy, Troy, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Ocean University Medical Center, Brick, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Southern Ocean County Medical Center, Manahawkin, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - The Cancer Institute at Saint Francis Hospital, East Hills, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Mount Sinai Chelsea, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Good Samaritan University Hospital, West Islip, New York
  - Atrium Health Stanly/LCI-Albemarle, Albemarle, North Carolina
  - Randolph Hospital, Asheboro, North Carolina
  - Messino Cancer Centers, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Levine Cancer Institute-SouthPark, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Levine Cancer Institute-Ballantyne, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Novant Health Cancer Institute - Kernersville, Kernersville, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - Novant Health Cancer Institute - Mount Airy, Mount Airy, North Carolina
  - Novant Health Cancer Institute - Wilkesboro, North Wilkesboro, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Novant Health Cancer Institute - Statesville, Statesville, North Carolina
  - Novant Health Cancer Institute - Thomasville, Thomasville, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Summa Health Medina Medical Center, Medina, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Cancer Treatment Centers of America, Tulsa, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Crozer-Keystone Regional Cancer Center at Broomall, Broomall, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Crozer Regional Cancer Center at Brinton Lake, Glen Mills, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Lancaster General Ann B Barshinger Cancer Institute, Lancaster, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Bryn Mawr Health Center, Newtown Square, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Eastern Regional Medical Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - The Radiation Oncology Center-Hilton Head/Bluffton, Hilton Head Island, South Carolina
  - Carolina Regional Cancer Center, Myrtle Beach, South Carolina
  - Rock Hill Radiation Therapy Center, Rock Hill, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - MD Anderson in The Woodlands, Conroe, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - Houston Methodist West Hospital, Houston, Texas
  - MD Anderson League City, League City, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - Houston Methodist Saint John Hospital, Nassau Bay, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Augusta Health Center for Cancer and Blood Disorders, Fishersville, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Japan (10):
  - Tohoku University School of Medicine, Sendai, Aoba-ku
  - Ehime University Hospital, Tōon, Ehime
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kagoshima City Hospital, Kagoshima, Kagoshima-ken
  - Gunma University Hospital, Gunma, Maebashi
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - Kyorin University Hospital, Mitaka-shi, Tokyo
  - Hiroshima University Hospital, Hiroshima
  - Shikoku Cancer Center, Matsuyama
  - Saitama Medical University International Medical Center, Saitama

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Higgins KA, Hu C, Ross HJ, Jabbour SK, Kozono DE, Owonikoko TK, Ritter TA, Williams TM, Welsh J, Simko JP, Movsas B, Xiao C, Kaira K, Gupta AK, Mohindra P, Dib EG, Brownstein J, Chun S, Kuzma CS, Kotecha R, Onitilo AA, Chen Y, Stinchcombe TE, Wang X, Paulus R, Bradley JD. Chemoradiation +/- Atezolizumab in Limited-Stage Small Cell Lung Cancer: Results of NRG Oncology/Alliance LU005. J Clin Oncol. 2026 Jan 13:JCO2501569. doi: 10.1200/JCO-25-01569. Online ahead of print. PMID 41529214
- [Derived] Higgins KA, Thomas A, Soto N, Paulus R, George TJ, Julian TB, Hartson Stine S, Markham MJ, Werner-Wasik M. Creating and Implementing a Principal Investigator Tool Kit for Enhancing Accrual to Late Phase Clinical Trials: Development and Usability Study. JMIR Cancer. 2022 Aug 25;8(3):e38514. doi: 10.2196/38514. PMID 36006678

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Chemotherapy, Radiation Therapy): Patients receive etoposide IV on days 1-3 and cisplatin IV or carboplatin IV on day 1. Cycles repeat every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo 3D-CRT or intensity-modulated radiation therapy (IMRT) twice daily (BID) for approximately 3 weeks or once daily (QD) for approximately 6-7 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo blood specimen collection throughout the trial.
Period: Overall Study
Arm/Group | Arm I (Chemotherapy, Radiation Therapy) | Arm II (Chemotherapy, Radiation Therapy, Atezolizumab)
Started | 270 | 274
Adverse Event Population ("As treated" randomized participants, counted on the arm matching the treatment they received.) | 257 | 264
Intent-to-treat (ITT) (Randomized participants counted on the treatment arm to which they were randomized) | 270 | 274
Completed (Participants contributing data to results are considered to have completed the study.) | 270 | 274
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Chemotherapy, Radiation Therapy) | Arm II (Chemotherapy, Radiation Therapy, Atezolizumab) | Total
Number analyzed (Participants) | 270 | 274 | 544
Age, Continuous [Median (Full Range); unit: years] | 67 [20 to 85] | 66 [44 to 84] | 66 [20 to 85]
Age, Customized [Count of Participants; unit: Participants]
  ≤ 49 | 11 | 5 | 16
  50 - 59 | 49 | 49 | 98
  60 - 69 | 115 | 127 | 242
  ≥ 70 | 95 | 93 | 188
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 140 | 277
  Male | 133 | 134 | 267
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 7 | 16
  Not Hispanic or Latino | 257 | 261 | 518
  Unknown or Not Reported | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 19 | 28 | 47
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 22 | 24 | 46
  White | 221 | 215 | 436
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 4 | 7 | 11
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — 0 = Asymptomatic; 1 = Symptomatic but completely ambulatory; 2 = Symptomatic, <50% in bed during the day; 3 = Symptomatic, >50% in bed, but not bedbound; 4 = Bedbound; 5 = Death
  Participants
    0 | 121 | 120 | 241
    1 | 136 | 142 | 278
    2 | 13 | 12 | 25
Platinum regimen (as randomized) [Count of Participants; unit: Participants]
  Carboplatin | 111 | 111 | 222
  Cisplatin | 159 | 163 | 322
RT Schedule (as randomized) [Count of Participants; unit: Participants]
  Twice a day (3 weeks) | 128 | 129 | 257
  Daily (6.5 weeks) | 142 | 145 | 287
T-Stage [Count of Participants; unit: Participants]
  T0 (No primary tumor) | 3 | 2 | 5
  T1 (Tumor ≤3 cm in size) | 96 | 89 | 185
  T2 (Tumor >3 cm but ≤5 cm or involves main bronchus, visceral pleura, or causes lung collapse.) | 58 | 60 | 118
  T3 (Tumor >5 cm but ≤7 cm or multiple tumors in the same lobe.) | 57 | 62 | 119
  T4 (Tumor >7 cm or invades nearby structures or has multiple tumors in different lobes.) | 46 | 52 | 98
  TX (Primary tumor cannot be assessed) | 10 | 9 | 19
N-Stage [Count of Participants; unit: Participants]
  N0: No regional lymph node involvement. | 20 | 26 | 46
  N1: Cancer in nearby lymph nodes. | 43 | 40 | 83
  N2: Cancer in lymph nodes in the center of the chest (mediastinum). | 147 | 148 | 295
  N3: Cancer in lymph nodes on the opposite side of the chest or above the collarbone. | 58 | 59 | 117
  NX: Cannot be assessed | 2 | 1 | 3
American Joint Committee on Cancer (AJCC) Stage [Count of Participants; unit: Participants] — The AJCC staging system is a standardized method for describing the extent and severity of cancer using the TMN System: T (Tumor): Size and extent of the primary tumor; N (Nodes): Involvement of regional lymph nodes; M (Metastasis): Presence of distant metastasis. Higher numbers indicate more advanced disease, zero indicates none. Categories may be further subdivided by letters, with higher letters indicating more advanced disease. The stage groupings are based on the TNM components, grouping cancers into stages (0-IV), with higher numbers indicating more advanced disease.
  Participants
    IA: T1, N0, M0 | 7 | 7 | 14
    IB: T2b, N0, M0 | 3 | 4 | 7
    IIA: T2b, N0, M0 | 2 | 4 | 6
    IIB: T1a-c or T2a-b, N1, M0; or T3, N0, M0. | 38 | 34 | 72
    IIIA: T1a-c or T2a-b, N2, M0; or T3, N1, M0; or T4, N0-1, M0. | 107 | 112 | 219
    IIIB: T1a-c or T2a-b, N3, M0; or T3, N2, M0; or T4, N2, M0. | 87 | 77 | 164
    IIIC: T3 or T4, N3, M0 | 26 | 36 | 62
Primary tumor location [Count of Participants; unit: Participants]
  Right Upper Lobe | 75 | 80 | 155
  Left Upper Lobe | 61 | 68 | 129
  Right Lower Lobe | 33 | 35 | 68
  Left Lower Lobe | 29 | 28 | 57
  Mediastinum | 20 | 19 | 39
  Other | 16 | 17 | 33
  Right Middle Lobe | 16 | 13 | 29
  Multiple Sites | 7 | 6 | 13
  Lingula | 4 | 5 | 9
  Carina | 4 | 1 | 5
  Main Bronchus, Left | 2 | 2 | 4
  Main Bronchus, Right | 2 | 0 | 2
  Undetectable Primary | 1 | 0 | 1
Forced Expiratory Volume in 1 second (FEV1) [Median (Full Range); unit: liters/second] — Forced expiratory volume (FEV1) is the amount of air one can forcefully exhale in one second after taking a deep breath, measured in liters per second. Population: Participants with data
  liters/second
    number analyzed (Participants) | 255 | 261 | 516
    (all) | 1.96 [0.42 to 6.08] | 1.99 [0.53 to 3.94] | 1.98 [0.42 to 6.08]
Percentage of Predicted FEV1 [Median (Full Range); unit: percentage of predicted value] — Percent predicted FEV1 expresses FEV1 as a percentage of the average FEV1 of a healthy person of the same age, sex, height, and ethnicity. Population: Participants with data
  percentage of predicted value
    number analyzed (Participants) | 255 | 263 | 518
    (all) | 71 [10 to 119] | 74 [23 to 123] | 72 [10 to 123]
Percentage of Predicted Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) [Median (Full Range); unit: percentage of predicted value] — DLCO measures how well a person's lungs transfers oxygen moves from the lungs into the bloodstream. Percent predicted DLCO expresses DLCO as a percentage of the average DLCO of a healthy person of the same age, sex, height, and ethnicity. Population: Participants with data
  percentage of predicted value
    number analyzed (Participants) | 248 | 257 | 505
    (all) | 67.5 [6.6 to 138] | 66 [12.7 to 138] | 66 [6.6 to 138]
Cigarette use [Count of Participants; unit: Participants]
  Current | 78 | 88 | 166
  Former | 185 | 181 | 366
  Never | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Survival rates and median survival time are estimated using the Kaplan-Meier method, censoring participants alive at time of analysis.
Time Frame: Randomization to date of death due or last follow-up. Median follow-up at the time of analysis was 23.8 months.
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Chemotherapy, Radiation Therapy) | Arm II (Chemotherapy, Radiation Therapy, Atezolizumab)
Number analyzed (Participants) | 270 | 274
months | 36.1 [28.1 to 42.5] | 31.1 [28.5 to 44.7]
Statistical Analysis 1: Comparison: Arm I (Chemotherapy, Radiation Therapy) vs Arm II (Chemotherapy, Radiation Therapy, Atezolizumab); Assuming exponentially distributed survival times, 480 eligible patients accrued uniformly over 48 months months) with 26 months additional follow-up after the last accrued patient would provide at least 85% power to detect a hazard ratio of 0.71 (median survival times of 38 months [Arm I] vs. 27 months [Arm II]) at a one-sided significance level of 0.025, after adjusting for type 1 error using group sequential methods for two interim analyses; Test type: Superiority; p = 0.5819, Log Rank; Stratified by radiation schedule (BID vs daily), chemotherapy (cisplatin vs carboplatin), and sex (male vs female). 1-sided significance level 0.025; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.82 to 1.34] — Stratified by radiation schedule (BID vs daily), chemotherapy (cisplatin vs carboplatin), and sex (male vs female). Reference level = Arm 1

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS failure event is defined as progressive disease (PD) determined by investigator per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or death due to any cause. PD is defined as at least a 20% increase in the sum of longest diameters of target lesions, and an absolute increase of at least 5 mm. The appearance of any new lesions is also considered progression. PFS rates and median PFS time are estimated using the Kaplan-Meier method, censoring participants alive without progression at the date of their last evaluable radiographic tumor assessment.
Time Frame: From randomization to progression or death due to any cause, whichever occurs first, or last tumor assessment if alive. MMedian follow-up at the time of analysis was 23.8 months.
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Chemotherapy, Radiation Therapy) | Arm II (Chemotherapy, Radiation Therapy, Atezolizumab)
Number analyzed (Participants) | 270 | 274
months | 11.4 [10.3 to 13.2] | 12.1 [10.9 to 15.2]
Statistical Analysis 1: Comparison: Arm I (Chemotherapy, Radiation Therapy) vs Arm II (Chemotherapy, Radiation Therapy, Atezolizumab); Test type: Superiority; Log Rank; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.80 to 1.21] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants by Highest Grade Adverse Event Reported
Description: Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grades adverse event severity as follows: 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, 5 = death related to adverse event. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data.
Time Frame: Randomization to last follow-up. Median follow-up at the time of analysis was 23.8 months.
Population: Adverse event population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Chemotherapy, Radiation Therapy) | Arm II (Chemotherapy, Radiation Therapy, Atezolizumab)
Number analyzed (Participants) | 257 | 264
Participants
  Overall: None reported | 4 | 0
  Overall: Grade 1 | 3 | 0
  Overall: Grade 2 | 8 | 9
  Overall: Grade 3 | 56 | 63
  Overall: Grade 4 | 182 | 168
  Overall: Grade 5 | 4 | 24
  Immune-mediated: None reported | 210 | 125
  Immune-mediated: Grade 1 | 19 | 29
  Immune-mediated: Grade 2 | 11 | 63
  Immune-mediated: Grade 3 | 14 | 31
  Immune-mediated: Grade 4 | 3 | 12
  Immune-mediated: Grade 5 | 0 | 4
  Non-Immune-Mediated: None reported | 4 | 0
  Non-Immune-Mediated: Grade 1 | 3 | 0
  Non-Immune-Mediated: Grade 2 | 8 | 10
  Non-Immune-Mediated: Grade 3 | 57 | 66
  Non-Immune-Mediated: Grade 4 | 181 | 168
  Non-Immune-Mediated: Grade 5 | 4 | 20

4. Secondary Outcome: Percentage of Participants With Confirmed Objective Response (Objective Response Rate (ORR))
Description: Objective response rate (ORR) is defined as the proportion of subjects whose best overall response (BOR) is a confirmed complete or partial response as determined by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 on two consecutive occasions ≥4 weeks apart.
Time Frame: Randomization to last radiographic tumor assessment. Median follow-up at the time of analysis was 23.8 months.
Population: Intent-to-treat population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Chemotherapy, Radiation Therapy) | Arm II (Chemotherapy, Radiation Therapy, Atezolizumab)
Number analyzed (Participants) | 270 | 274
percentage of participants | 59.6 [53.5 to 65.5] | 60.2 [54.2 to 66.1]

5. Secondary Outcome: Percentage of Participants With Local Progression
Description: Local progression is defined as intrathoracic tumor progression (failure in the lobe of the primary tumor or mediastinal lymph nodes) by RECIST 1.1 criteria determined by the investigator. Local progression rates are estimated by the cumulative incidence method, treating non-local progression (i.e., distant metastasis or failure in a different lung) and death without local progression as competing risks, and otherwise censoring participants alive at last tumor assessment. Treatment effect comparisons will utilize a cause-specific hazard function in which competing risks are censored.
Time Frame: From randomization to local progression, other progression, or death, whichever occurs first, or last tumor assessment if alive. Median follow-up at the time of analysis was 23.8 months. 1-, 2-, and 3-year rates are reported.
Population: Intent-to-treat population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Chemotherapy, Radiation Therapy) | Arm II (Chemotherapy, Radiation Therapy, Atezolizumab)
Number analyzed (Participants) | 270 | 274
percentage of participants
  1 year | 10.1 [6.6 to 14.4] | 8.1 [5.0 to 12.0]
  2 years | 14.3 [10.1 to 19.3] | 12.8 [8.8 to 17.5]
  3 years | 14.3 [10.1 to 19.3] | 12.8 [8.8 to 17.5]
Statistical Analysis 1: Comparison: Arm I (Chemotherapy, Radiation Therapy) vs Arm II (Chemotherapy, Radiation Therapy, Atezolizumab); Test type: Superiority; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.52 to 1.41] — Cause-specific hazard ratio stratified by radiation schedule (BID vs daily), chemotherapy (cisplatin vs carboplatin), and sex (male vs female). Reference level = Arm 1

6. Secondary Outcome: Distant Metastases-free Survival (DMFS)
Description: DMFS failure event is defined as first date of documented distant metastases (or failures in a different lung lobe) or death due to any cause, whichever occurs first. Participants with local progression prior to such an event are censored on the date of local progression. Participants with no post-baseline tumor assessment and alive at last follow-up are censored on the date of randomization. Participants alive without distant metastasis, failures in a different lung lobe, or local progression are censored on the date of their last evaluable radiographic tumor assessment. DMFS rates and median DMFS time are estimated using the Kaplan-Meier method.
Time Frame: Randomization to DMFS event or local progression, whichever occurs first, or last tumor assessment if alive. Median follow-up at the time of analysis was 23.8 months.
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Chemotherapy, Radiation Therapy) | Arm II (Chemotherapy, Radiation Therapy, Atezolizumab)
Number analyzed (Participants) | 270 | 274
months | 13.0 [11.3 to 18.2] | 16.8 [12.1 to 21.6]
Statistical Analysis 1: Comparison: Arm I (Chemotherapy, Radiation Therapy) vs Arm II (Chemotherapy, Radiation Therapy, Atezolizumab); Test type: Superiority; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.76 to 1.20] — Stratified by radiation schedule (BID vs daily), chemotherapy (cisplatin vs carboplatin), and sex (male vs female). Reference level = Arm I

7. Secondary Outcome: Percent of Participants With Deterioration in Functional Assessment of Cancer Therapy-Trial Outcome Index (FACT-TOI)
Description: FACT-TOI is a measure of 21 items that sums the functional well-being (FWB), physical well-being (PWB), and the lung cancer subscale (LCS) of the Functional Assessment of Cancer Therapy - Lung (FACT-L) quality of life (QOL) instrument. The FACT-TOI total score ranges from 0 to 84 with higher scores indicating better quality of life and functioning. Clinically meaningful decline is defined as a decrease from baseline of at least 5 points.
Time Frame: Baseline and 15 months after completion of chemoradiation (approximately 18 months after randomization)
Population: Intent-to-treat participants with FACT-TOI at baseline and 15 months after completion of chemoradiation (approximately 18 months after randomization).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Chemotherapy, Radiation Therapy) | Arm II (Chemotherapy, Radiation Therapy, Atezolizumab)
Number analyzed (Participants) | 102 | 110
Participants | 33 | 39

8. Secondary Outcome: Quality-adjusted Survival Months
Description: Quality-adjusted survival is calculated as the sum of weighted time intervals. Weight is the EuroQol 5-dimensional 5-level (EQ-5d-5L) index score, which measures health-related quality of life and ranges from 0 (death) to 1 (full health).
Time Frame: Baseline to death, last follow-up or two years, whichever occurs first.
Population: Eligible participants with baseline EQ-5D-5L index score and at least one follow-up EQ-5D-5L index score.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Arm I (Chemotherapy, Radiation Therapy) | Arm II (Chemotherapy, Radiation Therapy, Atezolizumab)
Number analyzed (Participants) | 174 | 180
months | 16.9 [16.1 to 17.7] | 17.3 [16.6 to 18.0]

9. Secondary Outcome: Change From Baseline in the 7 Item Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form Score
Description: The PROMIS fatigue score measures self-reported fatigue symptoms over the past 7 days. Possible scores range from 29.4 to 83.2, with higher scores indicating more fatigue. Change score is calculated by subtracting baseline from later score, with a positive change score indicating increased fatigue.
Time Frame: Baseline and 15 months after completion of chemoradiation (approximately 18 months after randomization)
Population: Intent-to-treat participants with score at baseline and 15 months after completion of chemoradiation (approximately 18 months after randomization).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Chemotherapy, Radiation Therapy) | Arm II (Chemotherapy, Radiation Therapy, Atezolizumab)
Number analyzed (Participants) | 102 | 111
score on a scale | -2.0 (9.9) | -1.9 (7.7)

10. Secondary Outcome: Molecular Subtyping
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2029-02

11. Other Pre Specified Outcome: Patient-reported Symptomatic Toxicities
Description: Will be measured by Patient Reported Outcomes - Common Terminology Criteria for Adverse Events (PRO-CTCAE). For each symptom and each domain (i.e., frequency, severity, and interference), counts and frequencies will be summarized for the worst score experienced by the patient by treatment arm.
Time Frame: Up to 15 months after completion of chemoradiation therapy
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Concordance Between Tumor and Circulating Cell Free Deoxyribonucleic Acid (cfDNA) Molecular Subtypes
Description: The concordance between molecular subtypes obtained via ribonucleic acid sequencing (RNAseq) on tumor tissue and methylation analysis on cfDNA will be assessed among patients who have both evaluable RNAseq and methylation results, where Cohen's Kappa and corresponding 95% confidence interval will be reported. In addition, the sensitivity and specificity of dichotomized cfDNA molecular subtypes (considering RNAseq as reference standard), along with the associated 95% confidence intervals, will be reported. Spearman rank correlation and associated 95% confidence intervals based on bootstrap between RNAseq and methylation will be reported.
Time Frame: Up to 5 years
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Treatment Effect by Sex
Description: Estimates of the primary outcome treatment effect and the corresponding 95% confidence intervals by sex will be provided.
Time Frame: Up to 5 years
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Treatment Effect by Race
Description: Estimates of the primary outcome treatment effect and the corresponding 95% CIs by race will be provided.
Time Frame: Up to 5 years
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Treatment Effect by Ethnicity
Description: Estimates of the primary outcome treatment effect and the corresponding 95% CIs by ethnicity will be provided.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline to the date of last known follow-up. Median follow-up was 23.8 months.
Description: All-cause mortality was assessed in the intent-to-treat population. Adverse events were assessed in adverse event population.
Arm/Group | Arm I (Chemotherapy, Radiation Therapy) | Arm II (Chemotherapy, Radiation Therapy, Atezolizumab)
All-Cause Mortality (participants affected / at risk) | 120/270 | 132/274
Serious Adverse Events (participants affected / at risk) | 106/257 | 159/264
Other Adverse Events (participants affected / at risk) | 253/257 | 263/264
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Chemotherapy, Radiation Therapy) (N=257) | Arm II (Chemotherapy, Radiation Therapy, Atezolizumab) (N=264)
Anemia (Blood and lymphatic system disorders) | 12 | 17
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 17 | 35
Hemolysis (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 6
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 4
Cardiac disorders - Other (Cardiac disorders) | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 4 | 2
Heart failure (Cardiac disorders) | 1 | 7
Myocardial infarction (Cardiac disorders) | 1 | 7
Myocarditis (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 2
Restrictive cardiomyopathy (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypophysitis (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Colitis (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 2 | 3
Diarrhea (Gastrointestinal disorders) | 3 | 7
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 4 | 2
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Esophageal pain (Gastrointestinal disorders) | 0 | 2
Esophageal stenosis (Gastrointestinal disorders) | 1 | 0
Esophageal ulcer (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 10 | 15
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 6 | 9
Oral pain (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 11
Death NOS (General disorders) | 2 | 2
Disease progression (General disorders) | 0 | 4
Fatigue (General disorders) | 0 | 5
Fever (General disorders) | 2 | 5
Flu like symptoms (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
General disorders and administration site conditions - Other (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 7
Pain (General disorders) | 1 | 1
Sudden death NOS (General disorders) | 0 | 2
Allergic reaction (Immune system disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 1
Bacteremia (Infections and infestations) | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 1
Bone infection (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 1 | 0
Encephalitis infection (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 2 | 4
Infections and infestations - Other (Infections and infestations) | 4 | 9
Lung infection (Infections and infestations) | 9 | 19
Meningitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 8 | 10
Skin infection (Infections and infestations) | 0 | 4
Stoma site infection (Infections and infestations) | 0 | 1
Thrush (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 4
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 3
Fracture (Injury, poisoning and procedural complications) | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 4
Blood bicarbonate decreased (Investigations) | 0 | 1
Cardiac troponin T increased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 0 | 3
Ejection fraction decreased (Investigations) | 0 | 1
INR increased (Investigations) | 0 | 1
Investigations - Other (Investigations) | 2 | 0
Lymphocyte count decreased (Investigations) | 5 | 4
Neutrophil count decreased (Investigations) | 28 | 27
Platelet count decreased (Investigations) | 18 | 11
Weight loss (Investigations) | 1 | 1
White blood cell decreased (Investigations) | 26 | 18
Anorexia (Metabolism and nutrition disorders) | 1 | 5
Dehydration (Metabolism and nutrition disorders) | 10 | 8
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 1
Hyponatremia (Metabolism and nutrition disorders) | 4 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 5
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 4
Headache (Nervous system disorders) | 1 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Nervous system disorders - Other (Nervous system disorders) | 1 | 0
Nystagmus (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Radiculitis (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 2 | 1
Somnolence (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 0 | 5
Syncope (Nervous system disorders) | 1 | 4
Transient ischemic attacks (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 2 | 6
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 | 0
Renal calculi (Renal and urinary disorders) | 2 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 12
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9 | 24
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 11
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 1
Arterial thromboembolism (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 2 | 12
Peripheral ischemia (Vascular disorders) | 0 | 2
Thromboembolic event (Vascular disorders) | 7 | 12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Chemotherapy, Radiation Therapy) (N=257) | Arm II (Chemotherapy, Radiation Therapy, Atezolizumab) (N=264)
Anemia (Blood and lymphatic system disorders) | 210 | 220
Febrile neutropenia (Blood and lymphatic system disorders) | 18 | 8
Palpitations (Cardiac disorders) | 12 | 24
Sinus tachycardia (Cardiac disorders) | 35 | 41
Tinnitus (Ear and labyrinth disorders) | 43 | 26
Hyperthyroidism (Endocrine disorders) | 1 | 36
Hypothyroidism (Endocrine disorders) | 8 | 49
Blurred vision (Eye disorders) | 33 | 41
Abdominal pain (Gastrointestinal disorders) | 28 | 35
Constipation (Gastrointestinal disorders) | 102 | 123
Diarrhea (Gastrointestinal disorders) | 59 | 101
Dry mouth (Gastrointestinal disorders) | 12 | 19
Dyspepsia (Gastrointestinal disorders) | 24 | 27
Dysphagia (Gastrointestinal disorders) | 98 | 86
Esophageal pain (Gastrointestinal disorders) | 17 | 17
Esophagitis (Gastrointestinal disorders) | 147 | 158
Gastroesophageal reflux disease (Gastrointestinal disorders) | 28 | 41
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 8 | 19
Mucositis oral (Gastrointestinal disorders) | 24 | 32
Nausea (Gastrointestinal disorders) | 139 | 165
Vomiting (Gastrointestinal disorders) | 68 | 72
Chills (General disorders) | 19 | 25
Edema limbs (General disorders) | 34 | 43
Fatigue (General disorders) | 182 | 200
Fever (General disorders) | 21 | 27
Malaise (General disorders) | 13 | 20
Non-cardiac chest pain (General disorders) | 28 | 40
Pain (General disorders) | 29 | 41
Infections and infestations - Other (Infections and infestations) | 12 | 27
Lung infection (Infections and infestations) | 14 | 27
Thrush (Infections and infestations) | 16 | 24
Upper respiratory infection (Infections and infestations) | 5 | 14
Urinary tract infection (Infections and infestations) | 18 | 12
Bruising (Injury, poisoning and procedural complications) | 8 | 14
Dermatitis radiation (Injury, poisoning and procedural complications) | 48 | 63
Fall (Injury, poisoning and procedural complications) | 15 | 20
Infusion related reaction (Injury, poisoning and procedural complications) | 8 | 15
Alanine aminotransferase increased (Investigations) | 25 | 44
Alkaline phosphatase increased (Investigations) | 29 | 59
Aspartate aminotransferase increased (Investigations) | 25 | 42
Blood bilirubin increased (Investigations) | 11 | 16
Creatinine increased (Investigations) | 45 | 59
Investigations - Other (Investigations) | 9 | 16
Lymphocyte count decreased (Investigations) | 163 | 172
Neutrophil count decreased (Investigations) | 220 | 226
Platelet count decreased (Investigations) | 189 | 212
Thyroid stimulating hormone increased (Investigations) | 7 | 15
Weight loss (Investigations) | 51 | 86
White blood cell decreased (Investigations) | 209 | 222
Anorexia (Metabolism and nutrition disorders) | 89 | 127
Dehydration (Metabolism and nutrition disorders) | 47 | 58
Hypercalcemia (Metabolism and nutrition disorders) | 9 | 14
Hyperglycemia (Metabolism and nutrition disorders) | 80 | 79
Hyperkalemia (Metabolism and nutrition disorders) | 16 | 30
Hypoalbuminemia (Metabolism and nutrition disorders) | 58 | 79
Hypocalcemia (Metabolism and nutrition disorders) | 38 | 58
Hypokalemia (Metabolism and nutrition disorders) | 71 | 95
Hypomagnesemia (Metabolism and nutrition disorders) | 60 | 71
Hyponatremia (Metabolism and nutrition disorders) | 85 | 102
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 26
Back pain (Musculoskeletal and connective tissue disorders) | 35 | 54
Chest wall pain (Musculoskeletal and connective tissue disorders) | 10 | 14
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 34 | 26
Muscle cramp (Musculoskeletal and connective tissue disorders) | 7 | 18
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 23
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 | 18
Dizziness (Nervous system disorders) | 80 | 97
Dysgeusia (Nervous system disorders) | 38 | 66
Headache (Nervous system disorders) | 57 | 85
Memory impairment (Nervous system disorders) | 19 | 33
Paresthesia (Nervous system disorders) | 9 | 15
Peripheral sensory neuropathy (Nervous system disorders) | 39 | 50
Tremor (Nervous system disorders) | 3 | 16
Anxiety (Psychiatric disorders) | 17 | 32
Depression (Psychiatric disorders) | 18 | 28
Insomnia (Psychiatric disorders) | 52 | 72
Cough (Respiratory, thoracic and mediastinal disorders) | 100 | 120
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 105 | 141
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 14
Hiccups (Respiratory, thoracic and mediastinal disorders) | 10 | 14
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 11 | 16
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 14
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 24 | 57
Productive cough (Respiratory, thoracic and mediastinal disorders) | 29 | 41
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 9 | 19
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 | 16
Sore throat (Respiratory, thoracic and mediastinal disorders) | 34 | 27
Wheezing (Respiratory, thoracic and mediastinal disorders) | 8 | 21
Alopecia (Skin and subcutaneous tissue disorders) | 80 | 75
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 26
Pruritus (Skin and subcutaneous tissue disorders) | 28 | 59
Rash acneiform (Skin and subcutaneous tissue disorders) | 6 | 16
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 21 | 51
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 7 | 26
Hypertension (Vascular disorders) | 53 | 41
Hypotension (Vascular disorders) | 28 | 43
Thromboembolic event (Vascular disorders) | 19 | 21

LIMITATIONS AND CAVEATS:
The second planned interim efficacy analysis met the early stopping rule for futility. Per the protocol, the second planned interim analysis occurred after 222 deaths had been reported across both arms combined. The final analysis would have otherwise taken place after 315 deaths.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/02/NCT03811002/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/02/NCT03811002/ICF_001.pdf